CLINICAL TRIAL: NCT03458741
Title: Regulation of Glycogen Supercompensation in Human Skeletal Muscle
Brief Title: How is Glycogen Supercompensation Regulated in Human Skeletal Muscle
Acronym: Supercomp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Janne Rasmuss Hingst, PhD, University of Copenhagen
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: Supercomp
Record Dates: First submitted 2018-02-15; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-03

CONDITIONS: Glycogen Depletion; Insulin Sensitivity
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Glycogen Supercompensation — The subjects arrived in the morning in the overnight fasted state at day 1, day 2 and day 5. Upon arrival in the morning the subjects were given a meal corresponding to 5% of their daily energy intake (~600-800 kJ). During the 5 day supercompensation regime the subjects were provided a predefined isocaloric diet containing 80% carbohydrates, 10% fat and 10% proteins. All food items were handle out to the subjects and compliance of the diet regime was ensured by survey.

SUMMARY:
Nine healthy, moderately fit male volunteers participated in the study. The subjects gave written informed consent after having been informed of any possible risk and discomfort associated with the study. The study was approved by the regional ethics committee in Denmark (Journal number: H-4-2013-071) and performed in accordance with the Declarations of Helsinki II.

All subjects underwent 3 clinical investigations (day 1, day 2 and day 5) during a 5 day glycogen supercompensation regime. The subjects were asked to refrain from physical activity and to eat a controlled diet containing 60% carbohydrates (CHO) for 4 days prior to the initial experiments.

Upon arrival at the laboratory on day 1, the subjects performed one-legged knee extensor exercise for 1 hour at 80% of PWL interspersed by 5 min bouts at 90% of PWL. This was followed by interval exercise until exhaustion containing 4 min bouts starting at 100% PWL followed by 1 min at 50% of PWL. Upon cessation of exercise the subjects showered and rested in the supine position for 4 hours. Then a 120 min hyperinsulinemic euglycemic clamp was initiated by a bolus insulin injection (9.0 mU/kg, Actrapid, Novo Nordisk, Denmark) followed by continuous insulin infusion (1.42 mU/kg/min insulin) reaching a level of plasma insulin around 100 µU/mL (n=9). At least 2 hours before the insulin clamp, catheters were placed in both femoral, one antecubital and one dorsal hand vein. A heat pad was placed around the lower part of the arm and hand in order to "arterialize" blood drawn from the hand vein. Substrate uptake/release across the legs was calculated by multiplying the arterial-venous (AV) difference in blood substrate concentration by femoral arterial blood flow (measured by ultrasound, Philips DICOM). Blood glucose levels were maintained at the euglycemic predefined target by continuously adjusting the glucose infusion rate (GIR) (20% glucose solution; Fresenius Kabi, Sweden). Concurrent measures of substrate AV differences and blood flow were performed every 20 min. Muscle biopsies from m. vastus lateralis were obtained under local anaesthesia (3-5 ml of Xylocaine, 20 mg/ml.) in the basal- and insulin-stimulated state (120 min) by use of needle biopsy technique. Muscle specimen were frozen within 20 sec in liquid nitrogen and stored at -80°C for further analysis. A new incision was made for every biopsy and spaced 4-5 cm apart.

This insulin clamp procedure in combination with basal and insulin stimulated muscle biopsies was repeated in the rested state (without prior exercise) on day 2 and day 5. The subjects arrived in the morning in the overnight fasted state at day 1, day 2 and day 5. During the 5 day supercompensation regime the subjects were provided a predefined isocaloric diet containing 80% carbohydrates, 10% fat and 10% proteins. All food items were handle out to the subjects and compliance of the diet regime was ensured by survey.

ELIGIBILITY:
Inclusion Criteria:

* male
* BMI between BMI 20-25 kg/m2
* healthy and not using medication
* not smoking
* habitual physical activity level of 2 - 6 hours pr. week
* no incidence of diabetes, cardiovascular disease or other metabolic diseases in close family

Exclusion Criteria:

* female
* BMI below 20 and above 25 kg/m2
* using medication
* smoking
* habitual physical activity level below 2 h pr. week or above 6 hours pr. week
* incidence of diabetes, cardiovascular disease or metabolic disease in close family

Ages: 25 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Insulin action in skeletal muscle | 1 week
  Insulin action in skeletal muscle was investigated during hyperinsulinemic euglycemic conditions by combining AV-difference with blood flow measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nutrition, Exercise and Sports, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No